CLINICAL TRIAL: NCT06911970
Title: Acute Effect of Moderate and High-Intensity Aerobic Exercise on the Anticancer Immune Response in Individuals Undergoing Treatment for Curable Cancer
Brief Title: Impact of Aerobic Exercise on the Anticancer Immune Response in Patients Receiving Cancer Treatment
Acronym: Immuno-Ex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-5606
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Breast Cancer; Non Metastatic Cancer
Keywords: cancer; exercise; T cells; NK cells; Migration; treatment; cytotoxic; immunology
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Each participant performed 2 experimental conditions (moderate continuous exercise and high-intensity interval exercise).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Condition HIIE (Experimental): Individuals undergoing cancer treatment will complete one session of high-intensity interval exercise (HIIE) with a ratio high-intensity/active recovery of 1 min /2 min. During the condition blood samples will be collected.
  Interventions: Other: Exercise
- Condition MOD (Active Comparator): Individuals undergoing cancer treatment will complete one moderate-intensity continuous exercise (MOD) session during which blood samples will be collected. MOD will consist of aerobic exercise that match external workload of HIIE.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Moderate-Intensity Continuous Exercise (MOD):
  The MOD condition will consist of a 37-minute continuous aerobic exercise session on ergocycle. This includes a warm-up and cool-down period at low intensity, and a 32-minute period at moderate intensity at a power corresponding to 50% of the last stop completed in the modified YMCA test completed in the preliminary visit.
  High-Intensity Interval Exercise (HIIE):
  The HIIE condition will consist of a 35-minute high-intensity aerobic exercise session on ergocycle. This includes a warm-up at low intensity, followed by 10 blocks of 1 minute at high intensity (110% of power highest poweroutput reached during the submaximal test) and 2 minutes of active rest (25% of highest power output).

SUMMARY:
The goal of this clinical trial is to determine to what extent anticancer immune cells mobilized by aerobic exercise exhibit migratory and functional capacity towards cancer cells in patients undergoing treatment for breast or colorectal cancer. The main questions it aims to answer are:

• Do anticancer immune cells mobilized by aerobic exercise will display migratory and functional capacity in patients undergoing treatment for curable breast or colorectal cancer?

Hypothesis: exercise will promote cell migration and these cells will display anti-cancer functional characteristics, suggesting a possible adjuvant and immunotherapeutic use of exercise.

• Do the magnitude of this anti-cancer immune response to exercise depend on the intensity of exercise?

Hypothesis: the achievement of a higher intensity of effort will enable greater mobilization of the cytotoxic lymphocytes of interest, but also the expression of markers predicting a more interesting adjuvant potential to immunotherapy.

Researchers will compare the effect of two exercise sessions, one moderate-intensity continuous exercise session (MOD) and one high-intensity interval exercise (HIIE) on the migration and anticancer potentials of mobilized immune cells.

Individuals aged between 40 and 70 with curable colon or breast cancer will be recruited to carry out a cross-over study with two experimental conditions. After a preliminary assessment visit, they will take part in:

* Two familiarization visits to validate the exercise prescription
* Two experimental visits (HIIE and MOD). During these conditions, blood samples will be taken before, after and 1 hour after the end of exercise to collect immune cells in the blood.

At the end of the visits, participants will leave with an accelerometer to wear for three days depending on conditions, and a notebook containing a questionnaire to assess fatigue levels over the same three days.

DETAILED DESCRIPTION:
In recent years, there has been growing interest in the therapeutic role of exercise in the context of oncology. Several murine models have demonstrated a reduction in tumor growth with aerobic exercise, which is partly due to the increased immunogenicity of the tumor microenvironment (TME). Aerobic exercise has the potential to mobilize cytotoxic immune cells, particularly those contributing to anticancer immunity (natural killer cells; NKc, and cytotoxic T lymphocytes; TCD8+), both in healthy individuals and in those living with cancer. In the latter, a session of aerobic exercise induces a transient rise in plasma lymphocytes, followed by their extravasation into inflamed tissues in the hours following exercise. This phenomenon, known as "exercise-immune-enhancement," appears to be heavily dependent on the adrenergic activation triggered by exercise. In other words, NKc and TCD8+ cells are mobilized in response to exercise of sufficient intensity, meaning a minimal physiological threshold must be reached during physical exertion, which should be identified on an individual basis (i.e., the second lactate threshold). However, it is crucial that cytotoxic immune cells mobilized by aerobic exercise can infiltrate the TME and exhibit characteristics that allow them to counter immune evasion mechanisms. Animal studies have shown that aerobic training increases the number of NKc and TCD8+ cells within primary tumors and delays tumor growth, supporting the hypothesis that exercise could stimulate tumor infiltration by cytotoxic lymphocytes acting within the TME. To date, no human studies conducted during treatment have confirmed this hypothesis.

The main objective of this study is to determine to what extent Tc and NK cells mobilized by aerobic exercise will exhibit migratory and functional capacity in patients undergoing treatment for curable breast or colorectal cancer. The secondary objective is to compare the effect of a moderate-intensity exercise (MOD) session with an high-intensity interval exercise (HIIE) session on the magnitude of this anti-cancer immune response to exercise and on the phenotypic and functional characteristics of the cells that have been mobilized.

The hypothesis is that exercise will promote cell migration, enhancing anti-cancer functionality, suggesting its potential as an adjuvant to immunotherapy. Additionally, higher exercise intensity is expected to increase mobilization of cytotoxic lymphocytes and expression of markers indicating stronger immunotherapeutic potential.

Forty-four individuals (aged 40-70) undergoing adjuvant treatment for breast or colorectal cancer will be recruited to participate in a randomized, crossover study with variable block size and counterbalanced design comparing the effect of two exercise modalities (MOD and HIIE), on the migratory and functional capacity of cytotoxic immune cells. An initial visit will be conducted to collect the following variables: resting heart rate and blood pressure, anthropometry, medical history, physical activity habits (questionnaire), gender identity, and aerobic capacity, which will be assessed using a submaximal graded exercise test on a cycle ergometer (modified YMCA). During MOD, participants will complete 32 minutes of cycling at 50% of the power output achieved during the last completed stage of the submaximal test. During the HIIE condition, participants will complete 10 intervals alternating 1 minute of intense effort at a power corresponding to 110% of the final stage completed in the modified YMCA test and 2 minutes of active recovery at 25% of the same stage, for a total duration of 30 minutes. Both experimental conditions are thus equivalent in terms of external effort load. During both exercise sessions, blood samples will be collected before, immediately after exercise cessation, and at 60 and 120 minutes post-exercise for complete blood counts and isolation of peripheral blood mononuclear cells (PBMCs) to assess migratory and functional capacity. Two familiarization sessions will precede the experimental conditions to test the respective prescriptions for MOD and HIIE to ensure that participants can complete the sessions at the required intensity to meet the research objective. A chemotactic gradient migration assay (Transwell assay) will be performed using the thawed PBMCs, and those that have migrated after 4 hours will be collected to characterize NKc and TCD8+ subpopulations and assess cytotoxicity potential using surface and intracellular antibody staining (fluorescence-activated cell sorting [FACS]).

The results of this study will help determine the extent to which the TCD8+ and NKc mobilized by aerobic exercise can migrate towards cancer cells, as well as the characteristics associated with anticancer cytotoxicity in individuals undergoing systemic treatment for curable breast or colorectal cancer. This data will help guide larger-scale randomized clinical studies with control groups aimed at confirming the adjuvant therapeutic role of individualized aerobic exercise in individuals undergoing systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-metastatic breast or colon cancer
* Age between 40 and 70
* Have started chemotherapy or immunotherapy treatment and have at least three treatments remaining in the cycle
* ECOG stage 0 to 1
* Be able to perform moderate-intensity aerobic exercise (MOD) or EPI type cycling according to the established prescription and without experiencing pain in connection with the bicycle saddle

Exclusion Criteria:

* Orthopedic, cardiac or metabolic limitation preventing safe aerobic exercise
* Non-controlled health condition
* Use of beta-blockers
* Planned surgery during the study period.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in migratory capacity of different peripheral blood mononuclear cells (Natural Killer Cells and T cells) | Before the start of the condition (t = 0 minute), at the end of the condition (t ≈ 35 minutes), 1 hour post-condition (t ≈ 95 minutes)
  Transwell migration assay
Change in the concentration and characterization of subpopulations of migrated peripheral blood mononuclear cells | Before the start of the condition (t = 0 minute), at the end of the condition (t ≈ 35 minutes), 1 hour post-condition (t ≈ 95 minutes)
  Flow cytometry

SECONDARY OUTCOMES:
Change in the concentration of inflammatory mediators in peripheral blood (chemokines, pro- and anti-inflammatory cytokines) | Before the start of the condition (t = 0 minute), at the end of the condition (t ≈ 35 minutes), 1 hour post-condition (t ≈ 95 minutes)
  Multiplex immunoassay
Change in catecholamines concentrations | Before the start of the condition (t = 0 minute), at the end of the condition (t ≈ 35 minutes), 1 hour post-condition (t ≈ 95 minutes)
  ELISA Kits
Cancer-Related Fatigue | During 3 days after the conditions.
  Multidimensional Fatigue Inventory 20 (MFI-20)
Changes in physical activity levels | During 3 days after the conditions
  Actigraph GT3X accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Eléonor Riesco, PhD, Principal Investigator — University of Sherbrooke, Faculty of Physical Activity Sciences, Department of Kinanthropology; Lee-Hwa Tai, PhD, Study Director — University of Sherbrooke, Faculty of Medicine and Health Sciences, Department of Immunology and Cellular Biology
Locations (1):
- Research Center on Aging, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No